CLINICAL TRIAL: NCT03191669
Title: Vaccine Exposure in Patients With Multiple Sclerosis in the Auvergne-Rhone-Alpes Region
Brief Title: Vaccine Exposure in Patients With MS
Acronym: Enquête Vaccin
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0169
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MS patients: Single group of patients with MS attending an outpatient MS clinic or hospitalization
  Interventions: Other: Auto-questionnaire

INTERVENTIONS:
Other: Auto-questionnaire — Single Auto-questionnaire administered during or after a consultation/hospitalization

SUMMARY:
Vaccines in MS patients have been controversial, in particular hepatitis B vaccine in the 90s and more recently human papillomavirus vaccine. There was an important flu incidence during the winter 2016-2017 that has revealed a low exposure to the flu vaccine in health professionals in France. Vaccine exposure of Multiple sclerosis (MS) patients has not been evaluated yet.

Objectives The primary objective is to evaluate exposure to the flu vaccine in patients with MS during the 2016-17 campaign. Secondary objectives are to evaluate exposure to mandatory vaccines, non mandatory vaccines, in the context of immunoactive treatments; to identify potential limitations to vaccines in general in patients with MS.

Methods Cross-sectional observational multicentric study, performed in Auvergne-Rhône-Alpes (France).

Data will be collected through an auto-questionnaire administered during an out-patient visit or hospitalization, during a two-week period.

Statistical analysis Description of the percentage of patients exposed to the flu vaccine, and to other vaccines. Stratification according to demographics (age, sex) and MS related criteria (disability level, relapse in the year before, disease-modifiying drug) Expected results Vaccine exposure of patients with MS will be put in perspective with the general population exposure. The study can provide information regarding potential reluctance of patients with MS towards vaccines. This could lead to develop specific communication tools for patients with MS and/or health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis according to MacDonald 2010 criteria
* Age 18 and more

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with MS attending an outpatient MS clinic or hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients exposed to seasonal flu vaccine in 2016-2017 | Two-weeks period in July 2017

CONTACTS AND LOCATIONS:
Overall Officials: Sandra VUKUSIC, Principal Investigator — Hôpital Neurologique Pierre Wertheimer - GHE
Locations (6):
- France (6):
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Service de Neurologie - Hôpital G. Montpied, Clermont-Ferrand
  - Service de Neurologie - CHU de Grenoble, Grenoble
  - Service de Neurologie - Hôpital Saint Joseph Saint Luc, Lyon
  - Cabinet de Neurologie - Clinique de la Sauvegarde, Lyon
  - Service de Neurologie - Hôpital Nord - CHU St Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No